CLINICAL TRIAL: NCT01971099
Title: Effects of Tribulus Terrestris in Women With Hypoactive Sexual Desire Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Selmo Geber, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TTM1
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Hypoactive Sexual Desire Disfunction
Keywords: sexual function; hypoactive; desire; androgens
MeSH Terms: conditions — Sedentary Behavior | interventions — Tribulus extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): patients will use placebo for 120 days
  Interventions: Other: Placebo
- Tribulus Terrestris (Experimental): patients will use Tribulus terrestris (750 mg/day) during 120 days
  Interventions: Drug: tribulus terrestris

INTERVENTIONS:
Drug: tribulus terrestris — patients will use 750mg/day of tribulus terrestris
  Other Names: tribulus
  Arms: Tribulus Terrestris
Other: Placebo — patients will take one pill a day (the same shape of the drug)
  Arms: Placebo

SUMMARY:
Hypoactive Sexual Desire Disorder (HSDD) is the most prevalent female sexual dysfunction in society and is strongly linked to the quality of life of women. The androgen hormones decline over age in the premenopausal period, which occurs around 20 years. Tribulus terrestris is a plant native to India, recommended in the treatment of infertility, low libido and impotence. Its main active ingredient is the protodioscin, which has been attributed to an increase in testosterone levels and improved sexual function. The aim of this study is to evaluate the effects of Tribulus Terrestris in premenopausal women with HSDD.

ELIGIBILITY:
Inclusion Criteria:

* regular menstrual cycle
* with no use of hormonal contraception within the last 3 months
* without any medication, drugs or alcohol.
* Healthy patients without systemic or psychiatric disease

Exclusion Criteria:

* Patients with amenorrhea and/or pregnant.

  * Patients who underwent bilateral oophorectomy.
  * Patient smoker (10 cigarettes per day).
  * Patients with blood pressure > 160/90 mm Hg.
  * Patient with breast or endometrial carcinoma.
  * Patients with a history of myocardial infarction.
  * Patient with Diabetes.
  * Patient with vaginal bleeding from any source.
  * Patients with hepatic injury.
  * Patients with active thrombophlebitis or thromboembolic disorders recent
  * Patients with interpersonal relationship problems with your relationship or partner
  * Patients with sexual problems from your partner

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Sexual Desire | 120 days
  we will use the "Quotient Sexual - Version Feminine (QS-F) brazilian questionary to make the evaluation

SECONDARY OUTCOMES:
serum levels of prolactin and thyroid-stimulating hormone (TSH) | 120 days
  blood test

OTHER OUTCOMES:
serum levels of testosterone and sex hormone-binding globulin (SHBG) | 120 days
  blood test

CONTACTS AND LOCATIONS:
Overall Officials: Selmo Geber, MD PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Hospital das Clinicas - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil